CLINICAL TRIAL: NCT00998452
Title: Dissemination of a Weight Management Program Among US Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0350
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2013-02

CONDITIONS: Body Weight
Keywords: Weight; Diet; Physical Activity; Veterans; MOVE! Program
MeSH Terms: conditions — Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOVE! (No Intervention): Participants will receive the usual VA MOVE! Program. These elements include a baseline assessment, brief clinic counseling session about weight, printed targeted health information on weight management and behaviors, and opportunities to participate in group sessions at the VA site and telephone follow-up from MOVE! clinic staff.
- MOVE*VETS (Active Comparator): Participants will receive the same MOVE! program as the control group plus 4 tailored newsletters on the study health behavior topics created from the baseline survey. Also 2-4 counseling calls from volunteer veteran peer counselors.
  Interventions: Behavioral: MOVE*VETS

INTERVENTIONS:
Behavioral: MOVE*VETS — Receiving 4 tailored newsletters on the study health behavior topics created from the baseline survey. Also 2-4 counseling calls from peer counselors.
  Arms: MOVE*VETS

SUMMARY:
This study is being conducted with the Veterans Affairs National Center for Health Promotion and Disease Prevention (VANCP), which is overseeing the current dissemination of MOVE! (Managing Overweight/Obesity for Veterans Everywhere), a national weight management program for veterans. It will be based at 10 local sites in the national network of VA medical settings and community-based outpatient clinics and will compare two different models for disseminating and implementing MOVE! using a randomized experimental design. One study arm will implement the MOVE* VETS! (Volunteer Education and Tailored Self-management and support) model that includes tailored newsletters and peer counseling MI calls and activities, and the other will receive the standard MOVE! program.

DETAILED DESCRIPTION:
The purpose of this research is to study the dissemination and implementation of MOVE!. MOVE! is a national weight management program for veterans that has moved form pilot to full dissemination. Overweight and obesity are rapidly rising in the United States and interventions to combat this epidemic are desperately needed. Within the VA population, approximately 70% of veterans are overweight and or obese. Participants will be male and female Veterans, aged 21 and over receiving health services at one of the 10 study sites, who qualify for the MOVE! program. We are recruiting a minimum of 800 -1000 Veterans to complete a baseline survey at the 10 VA sites participating in the study. Participants at the 10 VA sites are recruited during a primary care visit by primary care provider, they will not be chosen based on the presence or absence of any disease, thus health status will vary. The primary outcome measures will be participation after enrollment into MOVE! and participant weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Receiving primary care at the one of the 10 selected VA centers
* BMI 25 or over
* 21 years old, no upper age limit
* Pregnant women may participate in the study with the approval of the VA medical staff

Exclusion Criteria:

* Not a patient at one of the 10 VA sites
* BMI less than 25
* Under 21 years of age
* Pregnant without medical approval to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Primary study outcome measures at the participant level will be program participation and effectiveness in achieving weight loss. | At enrollment and 6 months post-enrollment

SECONDARY OUTCOMES:
Secondary outcome measures include improved self-management behaviors (diet and physical activity),psychosocial factors, awareness and utilization of program components/activities, and perceptions of the program/organization. | enrollment to 6 months post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Weiner, PhD, Principal Investigator — UNC Chapel Hill
Locations (11):
- United States (11):
  - West LA VAMC, West Los Angeles, California
  - West Haven VAMC, West Haven, Connecticut
  - Jesse Brown VAMC, Chicago, Illinois
  - Edward Hines Jr. VAMC, Hines, Illinois
  - Boston VAMC, Boston, Massachusetts
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Omaha VAMC, Omaha, Nebraska
  - Lineberger Comprehensive Cancer Center at UNC-CH, Chapel Hill, North Carolina
  - Audie L. Murphy VAMC, San Antonio, Texas
  - George E. Wahlen VAMC, Salt Lake City, Utah
  - VA Puget Sound HCS, Seattle, Washington